CLINICAL TRIAL: NCT00669279
Title: Non-Invasive Determination of Central Aortic Blood Pressure in Hypertensive Patients Treated With Controlled-Release Carvedilol or Atenolol
Brief Title: Effect of Carvedilol Controlled-Release (CR) and Atenolol on Central Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8COG11059
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Atenolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol CR (Experimental)
  Interventions: Drug: Carvedilol CR
- Atenolol (Experimental)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Carvedilol CR — Dose titration of 20mg by mouth once daily for 1 week, then 40mg by mouth once daily for 1 week, then 80mg by mouth once daily for 2 weeks
  Other Names: Coreg CR
  Arms: Carvedilol CR
Drug: Atenolol — Dose titration of 25mg by mouth once daily for 1 week, then 50mg by mouth once daily for 1 week, then 100mg by mouth once daily for 2 weeks
  Other Names: Tenormin
  Arms: Atenolol

SUMMARY:
The purpose of this research study is to determine whether atenolol or controlled release carvedilol lower blood pressure in the body as effectively as in the arm. Blood pressure measured in the aorta, a large blood vessel carrying blood away from the heart, may be a better measure of the harmful effects of high blood pressure on the body's organs. In the past, blood pressure has only been measured in the arms. However, blood pressure in the arms may not accurately reflect the blood pressure in the aorta and thus may mislead doctors treating high blood pressure. For this reason, we are testing whether two different medications for blood pressure, both in a class called beta blockers, have similar effects on blood pressure in the arm and aorta.

DETAILED DESCRIPTION:
Carvedilol reduces aortic wave reflection and improves left ventricular/vascular coupling: a comparison with atenolol (CENTRAL Study) is a prospective, open-label, comparative, randomized control trial that evaluated brachial and central hemodynamic profiles in patients taking atenolol or controlled-release carvedilol.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Hypertension (untreated or treated with no more then one anti-hypertensive drug)

Exclusion Criteria:

* Secondary forms of hypertension (including sleep apnea)
* Patients currently treated with two or more antihypertensive drugs
* Patients taking antihypertensive drugs with properly measured clinic systolic blood pressure greater then 170mmHg
* Isolated systolic hypertension
* Other diseases requiring treatment with blood pressure lowering medications
* Heart rate less then 55 beats/min (in the absence of beta-blocker therapy)
* Known cardiovascular disease including history of angina pectoris, heart failure, presence of a cardiac pacemaker, history of myocardial infarction or revascularization procedure, or cerebrovascular disease (including stroke and TIA)
* Known diabetes mellitus (Type 1 or 2)
* Renal insufficiency defined as a serum creatinine greater then 1.5mg/dL in males and 1.4mg/dL in females
* Primary renal disease
* Pregnancy or lactation
* History of Raynaud's syndrome
* Alcoholism and recreational drug use (due to compliance concerns)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Epstein, Pharm.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol CR: Controlled-release carvedilol 20 mg - Forced titration occurred in carvedilol to 40 mg at week one, and to 80 mg at week two.
- Atenolol: Atenolol 25 mg once daily - Forced titration occurred in atenolol to 50 mg at week one, and to 100 mg at week two.
Period: Overall Study
Arm/Group | Carvedilol CR | Atenolol
Started | 22 | 19
Completed | 22 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol CR | Atenolol | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.1) | 46.1 (9.9) | 46.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Central Aortic Blood Pressure
Time Frame: Measured at baseline and 4 weeks.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Carvedilol CR | Atenolol
Number analyzed (Participants) | 22 | 19
mmHg | -16.1 (10.4) | -16.0 (18.7)

2. Secondary Outcome: Peripheral Blood Pressure
Time Frame: Measured at baseline, 2 weeks, and 4 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Carvedilol CR | Atenolol
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

LIMITATIONS AND CAVEATS:
Small sample size, short duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No